CLINICAL TRIAL: NCT07101185
Title: Transition to Adulthood in People With Dystrophy: Social Cognition Mechanisms, Psychosocial Adjustment, and Mental Health and Coping Strategies.
Brief Title: Transition to Adulthood in People With Muscular Dystrophy
Acronym: TAMDY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Università di Padova Italy (Unknown); Fondazione Istituto Neurologico Nazionale Casimiro Mondino - IRCCS (Unknown); Istituto Giannina Gaslini - IRCCS (Unknown); Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other); Centro Clinico NeMO Ancona (Unknown); Fondazione Stella Maris - IRCCS (Unknown); Università degli Studi di Milano Statale (Unknown); Centro Clinico NeMO Brescia (Unknown); Fondazione Istituto Neurologico Carlo Besta - IRCCS (Unknown); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); I.R.C.C.S. Eugenio Medea - Associazione La Nostra Famiglia - Sede di Conegliano (Unknown); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Dipartimento di Neuroscienze Rita Levi Montalcini Torino (Unknown); Università Vita-Salute San Raffaele (Other); Università di Pisa (Unknown); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other); Associazione La Nostra Famiglia Eugenio Medea - Brindisi (Unknown); Scientific Institute, IRCCS E.Medea, Pasian di Prato (Unknown); Istituto delle Scienze Neurologiche di Bologna - IRCCS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Medea 152/24
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Duchenne / Becker Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; transition to adulthood,; social cognition; psychosocial adjustment; mental health and coping strategies
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Standardized neuropsychological measures of Theory of Mind will be also administered. The Virtual Reality (VR) scenario will be used to measure social cognition abilities in a subsample of 40 patients recruited at the centers of the Scientific Institute E. Medea in Bosisio and in Brindisi and at the Fondazione Mondino in Pavia, which have equipment and know-how for VR applications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm (Experimental): SOCIAL COGNITION- VIRTUAL REALITY
  Interventions: Device: VIRTUAL REALITY

INTERVENTIONS:
Device: VIRTUAL REALITY — The interventional part of the study is limited to 3 centers. It explores SOCIAL COGNITION throught a newly developed paradigm in Virtual Reality.
  In detail: an adapted version of the Virtual Reality Social Prediction Improvement and Rehabilitation Intensive Training (VR-SPIRIT) using a VR Head Mounted Display (HMD) will be implemented on a portable HMD, the Oculus Quest, equipped with two controllers with motion sensors that are used to track hand position.
  In a VR-SPIRIT session, participants are immersed in the playground scenario and engaged in a competition with four avatars. Each avatar has a pre-established probability to move toward one of the three described games.
  Different indices about a partecipant's performance are recorded automatically by the system during the session, such as the duration of each trial and the prediction score (percentage of trials in which the participant correctly predicted an avatar's intention).

SUMMARY:
The study will involve boys with Duchenne Muscular Dystrophy (DMD), from adolescence to adulthood living in Italy, and their families/ caregivers.

The Investigators want to explore patients' mental health, social cognition and perception of body image as well as patients'and caregivers' ability to adapt to changes related to both the disease and various personal and social needs, through the use of short and simple questionnaires, neuropsychological tests and neurocognitive evaluation in ecological scenarios using Virtual Reality. The desire for autonomy and the awareness of both personal and social difficulties in achieving them put a strain on both patients and their families.Some studies conducted in the USA and in various European countries underline that the transition to adulthood of patients with muscular dystrophy is featured by a good ability to adapt to the more advanced stages of the disease in general; nevertheless, facing the worsening of health entails experiences of anxiety and depression.In this historical phase, clinical trials of gene therapy and gene modulating therapies are involving an increasing number of patients, mainly represented by children in the early phase of the disease. Hence, adolescents and young adults could develop feelings of exclusion from research efforts, losing confidence and hope in any future improvement of their condition, social participation and quality of life.This study could lead to identify strengths and weaknesses in social cognition and psychosocial adaptation; through the evaluation of characteristics of patients/caregivers or exogenous factors influencing higher levels of social adaptation, we ultimately aim to define strategies to improve not only physical (already defined by guidelines) but also psychological care, social cognition and social support in all stages of DMD, particularly in later ones.

DETAILED DESCRIPTION:
In recent decades, various scientific studies have demonstrated the effectiveness of non-invasiveventilation therapy, steroid therapy and in the early setting of cardiologic therapy with the result of lengthening the life expectancy of DMD patients up to 30-40 years and more.These recent improvements in care open up new questions relating, on one hand, to the management of typical problems of adulthood such as independence, leaving the family of origin and the management of new health problems (physical and psychological), and, on other hand, the necessary acceptance that, despite the advances in research in the therapeutic field, at the moment most of older patients (or simply wheelchair bound ones) have no access or very low possibility to access to either experimental therapies or innovative treatments.The Investigators hypothesize from their clinical experience and from the few data reported in the literature that a more severe clinical involvement may be related in some patients, to an increase in anxiety and depression meanwhile in others the Investigators are witnessing a strengthening of life planning.Some preliminary activities aimed at improving the multidisciplinary care in the late stages of the disease have been suggested for DMD, but the Investigators are mainly focused on body care (cardiac, respiratory, anaesthetic, gastrointestinal, bone health care) (Quinlivan R 2021), whereas limited evidence has been collected and very few interventions have been implemented in the psychosocial sphere.In the Investigators' opinion, an exploration of the psychosocial adjustment, social cognition, coping strategies, body image and mental health in a wide population of Italian adolescents and young adults with DMD and their families is mandatory, with the aim to identify strengths and weaknesses in psychosocial adaptation and social cognition and to define possible ways of improving not only the physical (which is defined and revised in dedicated guidelines) but also the psychosocial care. According to the transactional stress and coping model, parents who cope with their children's condition through acceptance of the reality-rather than denial of it-and positive reinterpretation of the experience (e.g., finding of opportunities for growth), could have a better emotional regulation in the long term, with a positive influence on children's emotional well-being and mental health. Research is needed in teenagers and adults to evaluate the possibility to establish, reinforce and sustain the same virtuous cycle in the whole population of patients.Invetigators believe that interventions aimed at developing individual resilience may help to foster the well-being of persons with neuromuscular disorders and protect them from later severe psychopathology.

From clinical experience and from few studies reported in literature (Magliano 2013, Aho 2015, Gagliardi 1991, Pater 2023), each patients' response to potential stressors may be different and change over time suggesting different levels of psychosocial adaptation and coping strategies.The Investigators hypothesize to identify groups of patients with higher levels of psychosocial adaptation (and potentially lower risk of developing psychopathology), the analysis of the characteristics of these subjects and the identification of the factors playing a role in this positive attitude may be useful to define which personal and relational resources need to be supported or developed to improve quality of life; this could allow also prompts discussion with territorial authorities for greater consideration of these families and their needs (employment opportunities, accessible working spaces, recreational opportunities, etc.).

OBJECTIVES: The study therefore aims to:1) assess psychosocial adjustment, mental health and coping strategies through standardized measures in a large population of teenagers and adults with DMD and their caregivers;2) test social cognition mechanisms with standardized neuropsychological evaluation and newly-developed cognitive neuroscience paradigms that investigate emotional and social processing in ecological settings using Virtual reality in a subsample of patients;3) explore the body image perception and assess its impact on psychological well-being exploring the role of cognitive and motor impairment as possible mediators 4) investigate the interaction patterns between medical conditions, social cognition, psychosocial adjustment, mental health and coping strategies, in order to identify strengths to be supported and weaknesses to be reduced or counterbalanced. The project will ultimately pave the way for future development of cognitive and psychosocial interventions for improving psychosocial functioning and quality of life of the partecipants

ELIGIBILITY:
Inclusion Criteria:

* Defined diagnosis of DMD
* Age > 14 years
* Willingness and ability to comply to study procedures
* Comprehension of the study and Signature of the informed consent

Exclusion Criteria:

* Clinical history of cerebral palsy, severe intellectual deficit, severe behavioral disturbances
* absence of compliance to the studyof the patient and the caregivers.

Min Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
psychosocial adjustment, mental health and coping strategies | baseline visit
  To assess psychosocial adjustment, mental health and coping strategies through standardized measures in a large population of teenagers and adults with DMD and their caregivers
social cognition | baseline visit
  To test social cognition mechanisms with standardized neuropsychological evaluation and newly-developed cognitive neuroscience paradigms that investigate emotional and social processing in ecological settings using Virtual reality in a subsample of partecipants
body image | baseline visit
  To explore body image perception and assess its impact on psychological well-being exploring the role of cognitive and motor impairment as possible mediators
Correlation with medical conditions | baseline visit
  To investigate the interaction patterns between medical conditions and test on social cognition, psychosocial adjustment, mental health and coping strategies, to identify strengths to be supported and weaknesses to be reduced or counterbalanced.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Rare Disease- Rehabilitation Dept, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanzo' S, Tizzoni F, Previtali SC, Berardinelli A, Nobile M, Molteni M, Manzoni M, Tarabelloni A, Russo A, Delle Fave A, D'Angelo MG. Psychosocial resources and psychopathology among persons with neuromuscular disorders during the COVID-19 pandemic. BMC Psychol. 2024 Apr 29;12(1):243. doi: 10.1186/s40359-024-01742-5. PMID 38685111